CLINICAL TRIAL: NCT07104604
Title: Study on the Efficacy and Safety of Neoadjuvant Radiotherapy Combined With Toripalimab, Liposomal Irinotecan, and Capecitabine in the Treatment of pMMR Locally Advanced Rectal Adenocarcinoma With Low Rectal Involvement
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Affiliated Cancer Hospital of Shantou University Medical College (Other)
Responsible Party: Principal Investigator, Hao-Kai Hu, Clinical Professor，Doctor, Affiliated Cancer Hospital of Shantou University Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CancerShantouUMC 2
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Rectal Cancer
Keywords: Neoadjuvant therapy; rectal cancer; liposomal irinotecan; radiotherapy; immunotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — irinotecan sucrosofate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liposomal Irinotecan (Experimental): Treatment regimen:
  1. During radiotherapy: Radiotherapy 50Gy/25F + liposomal irinotecan 30mg/m² ivgtt qw w1-w4 + capecitabine 625mg/m² Bid, orally on radiotherapy days + tislelizumab 200mg ivgtt q3w;
  2. Radiotherapy-surgery interval: Liposomal irinotecan 70mg/m² ivgtt q3w + capecitabine 1000mg/m² Bid D1-D14 q3w + tislelizumab 200mg ivgtt q3w.
  Interventions: Drug: Liposomal Irinotecan

INTERVENTIONS:
Drug: Liposomal Irinotecan — In this study, the novel drug liposomal irinotecan was added, replacing the conventional formulation of irinotecan, and used as an intensified chemotherapy regimen (liposomal irinotecan + capecitabine) combined with immunotherapy and radiotherapy for neoadjuvant treatment of mid-lower rectal cancer.
  Other Names: New Neoadjuvant Treatment Approach

SUMMARY:
The goal of this clinical trial is to evaluating the efficacy and safety of radiotherapy combined with Tislelizumab, Liposomal Irinotecan, and Capecitabine in patients with locally advanced mid-lower rectal cancer with pMMR.. Patients would be included as:1. Aged between 18-75 years, with no gender restrictions; 2. Biopsy pathology confirmed as pMMR type locally advanced mid-lower rectal adenocarcinoma (tumor lower margin ≤ 10 cm from the anal verge); 3.With the following high-risk factors: T3N+/T4/N2/EMVI+/MRF+/lateral lymph node metastasis/inability to preserve anal function during surgery; 4. No distant metastasis observed in routine chest and abdominal CT scans.

ELIGIBILITY:
Here is the updated format for the **Eligibility Criteria** with bullet points for each item:

Inclusion Criteria:

* Age: 18-75 years, no gender restriction
* ECOG score 0-1
* Biopsy-confirmed pMMR (proficient mismatch repair) localized advanced low rectal adenocarcinoma (tumor's lower edge ≤ 10 cm from the anus)
* Presence of the following high-risk factors: T3N+/T4/N2/EMVI+/MRF+/lateral lymph node metastasis/inability to undergo sphincter-preserving surgery
* Routine chest and abdominal CT scans showing no distant metastasis
* Bone marrow function: Neutrophil count (ANC) ≥ 1.5 × 10^9/L, platelet count (PLT) ≥ 100 × 10^9/L, hemoglobin (Hb) ≥ 70 g/L
* Liver function: ALT, AST ≤ 2.5 × ULN (upper limit of normal); total bilirubin ≤ 1.5 × ULN; serum albumin ≥ 3 g/dL
* Kidney function: Serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance ≥ 60 ml/min (calculated using the Cockcroft-Gault formula)
* For females and patients with reproductive potential, a negative pregnancy test must be done within 72 hours before starting the treatment, and the patient must agree to avoid pregnancy during the study treatment and for 6 months after the treatment. For males with reproductive potential partners, the patient must agree to use adequate medically approved contraception during and for 90 days after the final study treatment
* Patients must agree to receive the study's neoadjuvant chemotherapy regimen and sign an informed consent form

Exclusion Criteria:

* Patients with a history of other malignancies within the past 5 years (except for cured and non-recurring cancers such as in situ carcinoma, basal cell carcinoma of the skin, etc.)
* Patients with active, uncontrolled bacterial, viral, or fungal infections requiring systemic treatment, defined by persistent signs/symptoms related to infection, which do not improve despite appropriate antibiotics, antiviral treatments, and/or other therapies
* Patients with uncontrolled systemic diseases, including unstable angina, myocardial infarction, congestive heart failure, severe unstable ventricular arrhythmia, history of severe pericardial disease, or other cardiovascular diseases; uncontrolled hypertension (defined as systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg despite appropriate antihypertensive treatment), or a history of hypertensive crisis, hypertensive encephalopathy; uncontrolled diabetes (fasting blood glucose ≥ 10 mmol/L), etc.
* Patients known to be allergic or intolerant to the treatment drugs or excipients used in this study
* Any clinical indicators showing contraindications to chemotherapy and surgery
* Patients using strong inhibitors or inducers of enzymes such as CYP3A4, CYP2C8, and UGT1A1
* Pregnant or breastfeeding women, and female patients of reproductive potential who refuse to use appropriate contraceptive measures during the study
* Patients who participated in other clinical trials within 4 weeks before enrollment
* Patients whom the investigator deems unsuitable for participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | 24 months
  Complete Remission Rate (CRR) refers to the percentage of patients who have achieved complete remission (CR) after treatment, typically in the context of cancer therapy. Complete remission means that all signs of cancer have disappeared, as determined by clinical, radiological, or pathological evaluation. However, this does not necessarily imply that the disease is cured, as microscopic cancer cells may still be present in the body and the patient may be at risk of relapse. CRR is an important measure used to assess the effectiveness of a treatment regimen, especially in clinical trials and cancer treatment protocols.The complete remission rate includes both pathological complete remission rate and clinical complete remission rate.

SECONDARY OUTCOMES:
Major Pathological Remission Rate | 24 months
  Major Pathological Remission Rate (MPRR) refers to the percentage of patients who achieve a significant reduction or near-total absence of tumor cells in pathological examination after receiving treatment. The threshold for defining "major" refers to a large proportion (e.g., ≥ 90%) of the tumor being eliminated or showing no viable malignant cells in the pathology report.

CONTACTS AND LOCATIONS:
Locations (1):
- Shantou University Medical College Cancer Hospital, Shantou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bang YJ, Li CP, Lee KH, Chiu CF, Park JO, Shan YS, Kim JS, Chen JS, Shim HJ, Rau KM, Choi HJ, Oh DY, Belanger B, Chen LT. Liposomal irinotecan in metastatic pancreatic adenocarcinoma in Asian patients: Subgroup analysis of the NAPOLI-1 study. Cancer Sci. 2020 Feb;111(2):513-527. doi: 10.1111/cas.14264. Epub 2019 Dec 20. PMID 31789476
- [Background] Wang-Gillam A, Li CP, Bodoky G, Dean A, Shan YS, Jameson G, Macarulla T, Lee KH, Cunningham D, Blanc JF, Hubner RA, Chiu CF, Schwartsmann G, Siveke JT, Braiteh F, Moyo V, Belanger B, Dhindsa N, Bayever E, Von Hoff DD, Chen LT; NAPOLI-1 Study Group. Nanoliposomal irinotecan with fluorouracil and folinic acid in metastatic pancreatic cancer after previous gemcitabine-based therapy (NAPOLI-1): a global, randomised, open-label, phase 3 trial. Lancet. 2016 Feb 6;387(10018):545-557. doi: 10.1016/S0140-6736(15)00986-1. Epub 2015 Nov 29. PMID 26615328
- [Background] Zhu J, Liu A, Sun X, Liu L, Zhu Y, Zhang T, Jia J, Tan S, Wu J, Wang X, Zhou J, Yang J, Zhang C, Zhang H, Zhao Y, Cai G, Zhang W, Xia F, Wan J, Zhang H, Shen L, Cai S, Zhang Z. Multicenter, Randomized, Phase III Trial of Neoadjuvant Chemoradiation With Capecitabine and Irinotecan Guided by UGT1A1 Status in Patients With Locally Advanced Rectal Cancer. J Clin Oncol. 2020 Dec 20;38(36):4231-4239. doi: 10.1200/JCO.20.01932. Epub 2020 Oct 29. PMID 33119477
- [Background] Yang Z, Gao J, Zheng J, Han J, Li A, Liu G, Sun Y, Zhang J, Chen G, Xu R, Zhang X, Liu Y, Bai Z, Deng W, He W, Yao H, Zhang Z. Efficacy and safety of PD-1 blockade plus long-course chemoradiotherapy in locally advanced rectal cancer (NECTAR): a multi-center phase 2 study. Signal Transduct Target Ther. 2024 Mar 11;9(1):56. doi: 10.1038/s41392-024-01762-y. PMID 38462629
- [Background] Rahma OE, Yothers G, Hong TS, Russell MM, You YN, Parker W, Jacobs SA, Colangelo LH, Lucas PC, Gollub MJ, Hall WA, Kachnic LA, Vijayvergia N, O'Rourke MA, Faller BA, Valicenti RK, Schefter TE, George S, Kainthla R, Stella PJ, Sigurdson E, Wolmark N, George TJ. Use of Total Neoadjuvant Therapy for Locally Advanced Rectal Cancer: Initial Results From the Pembrolizumab Arm of a Phase 2 Randomized Clinical Trial. JAMA Oncol. 2021 Aug 1;7(8):1225-1230. doi: 10.1001/jamaoncol.2021.1683. PMID 34196693